CLINICAL TRIAL: NCT05251896
Title: An Efficient Method of Eliminating M Protein in Patients With Multiple Myeloma by Plasma-free Replacement
Brief Title: Plasma-free Replacement in Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Fuling Zhou, Head,Division of Hematology; Professor of Hematology; Doctoral advisor, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00
Record Dates: First submitted 2021-11-23; First posted 2022-02-23 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cancer; Plasma exchange; Plasmapheresis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasma-free procedure (Experimental): Use albumin solution, lactated Ringer's solution, normal saline as replacement fluid
  Interventions: Procedure: Plasma-free procedure

INTERVENTIONS:
Procedure: Plasma-free procedure — Use albumin solution, lactated Ringer's solution, normal saline as replacement fluid

SUMMARY:
To evaluate whether the technique of no plasma exchange is suitable for the treatment, clinical efficacy, safety, and suitability of multiple myeloma patients with M protein abnormality or renal failure.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is the second most common hematological tumor after non-Hodgkin's lymphoma. The tumor cells originate from plasma cells in the blood pulp and are classified as plasma cells blood myeloma plasmacytomas by the WHO Tumor. It is characterized by abnormal proliferation of blood medullary plasma cells, accompanied by monoclonal immunoglobulin or light chain. Few patients are classified as non-secretory MM that does not secrete M protein. Multiple myeloma is often accompanied by multiple hemolytic damages, hypercalcemia, anemia, kidney damage, and a serious threat to the patients' lives, health, and quality of life, which have brought a heavy burden to society. Large amounts of M protein pass through the kidneys. At times, it causes acute or chronic renal failure; M protein interferes with the activity of coagulation factors, blocking platelet function, inducing bleeding; and a large amount of M protein can also lead to hyperviscosity syndrome, increase circulatory resistance, and small blood vessel thrombosis Plug, cause various neurological diseases such as blindness, and further aggravate the progression of kidney injury. Patients with hematological myeloma nephropathy already existed at the time of diagnosis, severe patients may die due to renal insufficiency, so the patient was removed immunity globulin in the body to improve the signs of hyperviscosity and clinical symptoms is the focus of clinical research.

In this study, on the basis of previous studies, albumin-free plasma exchange fluid treatment was given to analyze the effects of clinical symptoms, erythrocyte sedimentation rate, blood routine, albumin, renal function, calcium content, and immunoglobulin.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of MM 2. A stable condition after routine treatment 3. Clinical diagnosis of renal insufficiency or M protein abnormalities 4．more than 18 years old 5．With liver and kidney function 6. With normal heart function; 7. Physical condition score 0-2 (ECOG score) 8. Get informed consent from the patient or family member.

Exclusion Criteria:

1. Allergies or obvious contraindications to any drug;
2. Myocardial infarction and cardiac insufficiency
3. Other malignant tumors
4. TB patients and HIV positive patients 5．Other blood system diseases

6. Pregnant or lactating women; 7. Not understand or follow the protocol; 8. Allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change from M protein content in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  M protein content in plasma
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  WBC
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  RBC
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  PLT
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  Hb
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  Sodium ion
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  Potassium ion
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  eGFR
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  Creatine
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  β2-MG
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  UA
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  ALB
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  GLB
Adverse event: Low blood pressure | Day 1
  Low blood pressure
Adverse event: | Day 1
  Headache
Adverse event: Difficulty breathing | Day 1
  Difficulty breathing
Adverse event: Numbness | Day 1
  Numbness

SECONDARY OUTCOMES:
Safety and Tolerability Assess patient symptoms | Day 0，Day 1
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Fuling Zhou, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China